CLINICAL TRIAL: NCT03441932
Title: Evaluation of Morbidity and Mortality Associated With Dysphagia in Stroke Patients Based on Pharyngeal Residue Severity: A Prospective Study
Brief Title: Evaluation of Morbidity and Mortality Associated With Dysphagia in Stroke Patients Based on Pharyngeal Residue Severity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SaintJU
Record Dates: First submitted 2018-01-18; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Dysphagia Following Cerebral Infarction
Keywords: Dysphagia; Pharyngeal residue scale; Stroke; Pneumonia
MeSH Terms: conditions — Deglutition Disorders; Stroke; Pneumonia

STUDY DESIGN:
Intervention Model Description: * Dysphagia screening in the Emergency department for any patient admitted to Hotêl-Dieu de France university hospital for Stroke based on the " Emergency department dysphagia-screening tool".
  * Subjets will be then sorted in two groups:
  > 1-Screening passed > 2-Screening failed
  • Subjets within the two groups will after than have FEES with videotaping of pharyngeal phase after giving subjects a standardised food consisting of "thin Puree". An ENT resident blinded to the result of the screening test will do this intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dysphagia screening failed arm (Active Comparator): Subjets within the this arm will have FEES with videotaping of pharyngeal phase after giving subjects a standardised food consisting of "thin Puree". An ENT resident blinded to the result of the screening test will do this intervention
  Interventions: Procedure: Fiberoptic endoscopic evaluation of swallowing (FEES)
- Dysphagia screening passed arm (Active Comparator): Subjets within the this arm will have FEES with videotaping of pharyngeal phase after giving subjects a standardised food consisting of "thin Puree". An ENT resident blinded to the result of the screening test will do this intervention
  Interventions: Procedure: Fiberoptic endoscopic evaluation of swallowing (FEES)

INTERVENTIONS:
Procedure: Fiberoptic endoscopic evaluation of swallowing (FEES) — Subjets within the two groups will after than have FEES with videotaping of pharyngeal phase after giving subjects a standardised food consisting of "thin Puree".

SUMMARY:
Specific objectives:

* Evaluation of morbidity and mortality associated with the severity of pharyngeal residue in patients admitted to Hotêl-Dieu de France university hospital for Stroke based on the "The Yale pharyngeal residue scale"
* Evaluation of the accuracy of screening protocol of Dysphagia at the Emergency Department in patients admitted for stoke based on the "Emergency Department Dysphagia Screening Tool"

DETAILED DESCRIPTION:
Dysphagia after stroke is common, affecting 27% to 64% of patients. Complications of dysphagia include aspiration leading to chest infection and pneumonia, malnutrition, inability to rehabilitate, increased risk of infection, prolonged length of stay in hospital, and an increased risk of death.

Deglutologists who use FEES have long lamented the fact that there was no reliable, validated, anatomically defined, image-based, and easily used pharyngeal residue severity rating scale. All that one had to rely on was the "impression" of residue severity, the definition of which varied from endoscopist to endoscopist In order for any scale to gain widespread acceptance, it must be user friendly, easy to learn, reliable to interpret, and generalizable to all patients undergoing FEES. Such a scale now exists, and it is the Yale Pharyngeal Residue Severity Rating Scale

Need for a trial: The relation between the severity of the pharyngeal residue and the risk of aspiration and subsequently the morbidity and mortality in stroke patients is not well defined yet.

Thus, the purpose of this study was to determine the morbidity and mortality associated with the severity of pharyngeal residue in a specific population: stroke patients

Another objective of the study is to evaluate the accuracy of Emergency department (ED) dysphagia screening in stroke patients compared to a standard swallowing evaluation with FEES.

All patients admitted to Hotêl-Dieu de France university hospital for stroke will be evaluated for dysphagia using the ED dysphagia-screening tool. Preliminary data on the accuracy of the "ED dysphagia screening tool" are promising (Sensitivity of 96%)

In this study outcomes between 2 groups will be evaluated; (ED failed screening group and ED Screening passed group) and thus be able to validate results of previous studies concerning sensitivity and accuracy of the screening tool mentioned previously and finally to be able to identify stroke patients eligible for early oral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients admitted for Stroke (Ischemic or hemorragic)
* Patients reachable by phone call

Exclusion Criteria:

* Previous history of major head and neck surgery
* Previous or actual history of treatment by chemotherapy or radiotherapy for a head and neck neoplasm
* Current Head and neck neoplasm
* Previous or current history of esophageal carcinoma
* Esophageal motility disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
incidence of Aspiration pnemonia | From date of inclusion till 1 year post inclusion in the study
  Evaluation of aspiration pneumonia risk associated with the severity of pharyngeal residue in patients admitted to Hotêl-Dieu de France university hospital for Stroke based on the "The Yale pharyngeal residue scale".
  The Yale Pharyngeal Residue Severity Rating Scale can be used for both clinical advantages and research opportunities.
  Clinically, clinicians can now accurately classify vallecula and pyriform sinus residue severity as none, trace, mild, moderate, or severe for diagnostic purposes, determination of functional therapeutic change, and evaluation of prognosis

CONTACTS AND LOCATIONS:
Overall Officials: HUSEIN SMAYLI, M.D, Principal Investigator — Hotêl-Dieu de France university hospital, Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner-Lawrence DE, Peebles M, Price MF, Singh SJ, Asimos AW. A feasibility study of the sensitivity of emergency physician Dysphagia screening in acute stroke patients. Ann Emerg Med. 2009 Sep;54(3):344-8, 348.e1. doi: 10.1016/j.annemergmed.2009.03.007. Epub 2009 Apr 11. PMID 19362752
- [Result] Neubauer PD, Hersey DP, Leder SB. Pharyngeal Residue Severity Rating Scales Based on Fiberoptic Endoscopic Evaluation of Swallowing: A Systematic Review. Dysphagia. 2016 Jun;31(3):352-9. doi: 10.1007/s00455-015-9682-6. Epub 2016 Jan 11. PMID 26753927